CLINICAL TRIAL: NCT01347541
Title: Piloting Acute Care to Primary Care Linkage of Safety Net Patients
Acronym: TSOS III
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Inadequate recruitment
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Douglas Zatzick, Professor, University of Washington
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 40069
Record Dates: First submitted 2011-04-29; First posted 2011-05-04 (Estimated); Results first posted 2021-02-11 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-02

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Cognitive Behavioral Therapy; Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stepped care (Experimental): Combination of behavioral therapy and drug therapy
  Interventions: Behavioral: Cognitive Behavioral Therapy; Behavioral: Motivational Interviewing; Drug: FDA-Approved Anti-Anxiety Medications
- Standard care provided to injured trauma survivors (Active Comparator)
  Interventions: Behavioral: Standard Care Control

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Behavioral therapy includes standard cognitive behavioral therapy, with an emphasis on behavioral activation. Treatment is administered on the basis of the participants' individual needs and may continue for up to 12 months.
  Other Names: CBT
  Arms: Stepped care
Behavioral: Motivational Interviewing — Motivational interviewing is designed to address alcohol and drug use.
  Other Names: MI
  Arms: Stepped care
Drug: FDA-Approved Anti-Anxiety Medications — Participants assigned to receive the combination therapy may receive one or more of the following medications based on their individual needs: fluoxetine, sertraline, paroxetine, buspirone, propranolol, trazodone, and any of the benzodiazepines. Participants may begin receiving medication immediately or anytime within the 12 months post-injury. Form, dosage, frequency, and duration depend on patient need, but all are prescribed in accordance with standards of care.
  Arms: Stepped care
Behavioral: Standard Care Control — Standard care control includes the usual treatment for injured trauma survivors
  Other Names: BA
  Arms: Standard care provided to injured trauma survivors

SUMMARY:
This pilot study will evaluate the implementation of a stepped care intervention that combines Cognitive-Behavioral Therapy, Motivational Interviewing, psychotropic medications, and information technology innovations at a level 1 trauma center to community linkage components to reduce the symptoms of posttraumatic stress disorder and related comorbidities in injured trauma survivors treated in the emergency department and surgical inpatient settings.

DETAILED DESCRIPTION:
The investigators plan to implement a pilot linkage program in which trauma center based care facilitators will use a population-based recruitment strategy to facilitate outpatient follow-up for acutely injured trauma center inpatients and emergency department patients. All patients recruited into the trial will be low income patients with one or more of the following characteristics: being uninsured, low income older adults, low income mothers, and other high risk individuals who lack health insurance. Patients will be linked for care to one of the community health centers participating in Washington State.

In phase I, patients will be recruited from the trauma center inpatient trauma surgery service and emergency departments. In phase one, no randomization will occur; patients will be linked to one of the community health centers. Patients who consent to the protocol will be assessed in the surgical inpatient units or emergency department. After the baseline assessment, all patients will be immediately assigned a bachelor's, MSW, or RN level care manager. The care managers will elicit and address posttraumatic concerns, and attempt linkage of patients to community programs. Care managers may also deliver motivational interviewing and cognitive behavioral therapy interventions. Patient may also be linked to psychopharmacologic interventions targeting PTSD. Follow-up assessments will occur in the weeks and months after the injury and will assess patterns of health service utilization and symptomatic outcomes. Phase I will establish the feasibility of recruitment and follow-up, acceptability of care management for patients, as well as the pragmatics of linkage to community programs.

Piloting in phase II will depend on the results of phase I; the phase II pilot will build and extend upon phase I. In phase II, patients will be randomized to either intervention or control conditions. Patients randomized to the intervention condition will be met by a care manager who may address patients' initial needs and concerns. Care managers may also deliver Motivational Interviewing and Cognitive Behavioral Therapy interventions. Patients may also be linked to psychopharmacologic interventions targeting PTSD. The care manager will attempt to link patients to participating community health centers. Linkages may occur by the telephone, or through web-based clinical registry tools that are under development by the intervention team. Some linkages may occur in person. To determine if intervention patients are successfully linked more frequently than controls, all patients will be followed from the time of designation at hospital admission to outpatient primary care appointments. Follow-up outcome assessments will occur in the weeks and months post-injury and will includes assessments of patterns of health service utilization, function, and symptomatic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Admitted to Harborview Medical Center with injuries sufficiently severe enough to require inpatient admission
* Experienced a traumatic injury
* Exhibits symptoms of PTSD while in the hospital ward
* Low-income

Exclusion Criteria:

* History of head, spinal, or other injury that may prevent participation in the ward interview
* Requires immediate intervention due to conditions such as self-inflicted injury, active psychosis, or active mania
* Currently incarcerated
* Likely to face criminal charges
* Lives outside of the state of Washington
* Not low-income

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Zatzick, MD, Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States

REFERENCES:
- [Background] Zatzick DF, Roy-Byrne P, Russo JE, Rivara FP, Koike A, Jurkovich GJ, Katon W. Collaborative interventions for physically injured trauma survivors: a pilot randomized effectiveness trial. Gen Hosp Psychiatry. 2001 May-Jun;23(3):114-23. doi: 10.1016/s0163-8343(01)00140-2. PMID 11427243
- [Background] Zatzick D, Roy-Byrne P, Russo J, Rivara F, Droesch R, Wagner A, Dunn C, Jurkovich G, Uehara E, Katon W. A randomized effectiveness trial of stepped collaborative care for acutely injured trauma survivors. Arch Gen Psychiatry. 2004 May;61(5):498-506. doi: 10.1001/archpsyc.61.5.498. PMID 15123495

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stepped Care | Standard Care Provided to Injured Trauma Survivors
Started | 3 | 1
Completed | 3 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stepped Care | Standard Care Provided to Injured Trauma Survivors | Total
Number analyzed (Participants) | 3 | 1 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.33 (18.01) | 31 (NA) — Only one patient was recruited into the control arm, so standard deviation cannot be calculated. | 35.75 (15.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 0 | 1
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Alcohol Use Disorders Identification at 1 Month
Description: The investigators will use the Alcohol Use Disorders Identification Test (AUDIT) as a continuous measure. The 10-item scale score ranges from 0-40, with higher values indicating a worse outcome.
Time Frame: Baseline, Up to 12 months after injury
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Stepped Care | Standard Care Provided to Injured Trauma Survivors
Number analyzed (Participants) | 3 | 1
score on a scale | -1.7 [-7.9 to 4.6] | -2.0 [NA to NA] — Only one participant was recruited for the standard care arm of this pilot, so no confidence interval can be calculated.

2. Primary Outcome: Change From Baseline PTSD Checklist Civilian (PCL-C) at 1 Month
Description: The investigators will use the PTSD Checklist - Civilian (PCL-C). The scoring of the scale ranges from a minimum of 17 to a maximum of 85, with higher scores indicating a worse outcome. The measure can also provide a rating of symptoms consistent with a diagnosis of PTSD.
Time Frame: Baseline, Up to 12 months after injury
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Stepped Care | Standard Care Provided to Injured Trauma Survivors
Number analyzed (Participants) | 3 | 1
score on a scale | -4.0 [-55.3 to 47.3] | -14.0 [NA to NA] — Only one participant was recruited for the standard care arm of this pilot, so no confidence interval can be calculated.

3. Primary Outcome: Change in Functional Status at 1 Month
Description: The investigators will use the Medical Outcomes Study Short Form healthy survey (MOS SF-12/36) physical components summary to assess physical function. The minimum and maximum scores are 0-100 with higher scores representing a better outcome.
Time Frame: Baseline, Up to 12 months after injury
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Stepped Care | Standard Care Provided to Injured Trauma Survivors
Number analyzed (Participants) | 3 | 1
score on a scale | -1.9 [-11.5 to 7.8] | 4.0 [NA to NA] — Only one participant was recruited for the standard care arm of this pilot, so no confidence interval can be calculated.

4. Secondary Outcome: Increased Satisfaction With Global Care
Description: Assessed using the Posttraumatic Growth Inventory (PTGI) and Satisfaction with Care (NSCOT)
Time Frame: Up to 12 months after injury
Population: Data were not collected
Arm/Group | Stepped Care | Standard Care Provided to Injured Trauma Survivors
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Injury Relapse
Description: Assessed using Healthcare Utilization Questions (NSCOT)
Time Frame: Up to 5 years after injury
Population: Data were not collected
Arm/Group | Stepped Care | Standard Care Provided to Injured Trauma Survivors
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Work, Disability, and Legal Outcomes
Description: Assessed using Work, Disability and Legal (NSCOT) and Sheehan Disability Scale (SDS)
Time Frame: Up to 12 months after injury
Population: Data were not collected
Arm/Group | Stepped Care | Standard Care Provided to Injured Trauma Survivors
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Stepped Care | Standard Care Provided to Injured Trauma Survivors
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/1
Other Adverse Events (participants affected / at risk) | 0/3 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No